CLINICAL TRIAL: NCT04189471
Title: Recovery After Cerebral Hemorrhage--Improving Outcomes for Patients With Life-Threatening Neurologic Illness
Brief Title: Improving Outcomes for Patients With Life-Threatening Neurologic Illness
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Gunjan Parikh, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00056063
Record Dates: First submitted 2019-07-30; First posted 2019-12-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Intraventricular Hemorrhage; Nontraumatic Haemorrhage; Status Epilepticus
Keywords: hemorrhage; intracerebral hemorrhage; SAH; Nontraumatic Haemorrhage; ICH; subarachnoid hemorrhage; status epilepticus
MeSH Terms: conditions — Cerebral Hemorrhage; Subarachnoid Hemorrhage; Status Epilepticus; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — 12 mL of blood to be collected for RNA, DNA, and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

While the intensive care of patients with life-threatening brain illnesses has advanced tremendously, a large number of therapies are still without proper scientific support.

This can be partly explained by the fact that mechanisms of initial brain injury are still not well understood. Why additional neurological injury occurs during a patient's stay in the NeuroCritical Care Unit (NCCU) despite current best, evidence-based clinical practices, is also not well understood. However, over the past decade, better tools have become available to measure and monitor the impact of our clinical care on the rapidly changing physiology and chemistry of the injured brain. Some of these tools are CT, MRI, ultrasound, and catheter-based technology measuring blood flow and metabolism. These tools have enabled earlier detection of injury and complications and newer therapeutic strategies.

Purpose:

Examine disease pathways common to all brain injuries seen in the University of Maryland's 22-bed NCCU. Life-threatening neurological illnesses cared for in the NCCU include massive stroke, bleeding in and around the brain (subarachnoid hemorrhage, intracerebral hemorrhage, subdural hemorrhage, intraventricular hemorrhage), brain tumors, difficult to control seizures, neurologic infections, nerve and muscle diseases (such as myasthenia gravis or Guillain-Barre Syndrome), and spinal cord disorders among others. Many NCCU patients are comatose or paralyzed and may suffer injuries in other parts of the body as well.

This effort will require the creation of a robust clinical database for the capture of data including patient characteristics (age, sex), clinical characteristics, medical treatments, surgical interventions, physiological data (such as vital signs, cerebral blood flow, intracranial pressure, cerebral oximetry, etc), laboratory data, and standard-of-care diagnostic studies such as electroencephalography (EEG), ultrasound, CT, MRI, and angiograms. Similar databases exist at other major centers for neurocritical care and have been instrumental to the identification of characteristics both predictive of and associated with outcomes of patients long after their stay in the NCCU.

In addition, the samples collected will be included in the University of Maryland Medicine (UMM) Biorepository which is a shared resource to enable biomedical research by University of Maryland faculty.

DETAILED DESCRIPTION:
The objective of the proposed minimal-risk, non-interventional retrospective (January 2012 onwards) as well as prospective, cross-sectional observational study (i.e., NCCU Research Repository) is to better understand the common pathophysiological pathways of life-threatening neurological illnesses, examine how systemic complications (e.g., fever, hyperglycemia, undernutrition, and infections) and our standard-of care management of them may exacerbate brain injury, and determine the impact of injury and intervention on functionally-relevant outcomes.

A systematically collected cohort may have an especially important role in the NCCU where RCTs are difficult to implement or may lack generalizability, and wherein there are pitfalls in research derived solely from administrative databases. This relational database will capture all patients admitted to University of Maryland's dedicated 22-bed adult NCCU. The investigators will not initially collect all potentially relevant fields unique to specific diagnoses. However, future disease-specific studies will allow the addition of data fields in this flexible database environment. This approach will include the tiered acquisition of patient characteristics (age, sex), clinical characteristics, standard-of-care medical treatments and surgical interventions, physiological data (such as vital signs, cerebral blood flow, intracranial pressure, cerebral oximetry etc), laboratory data, and diagnostic studies--particularly neurophysiology, neuropathology, and neuroimaging. Some data elements are inherently less reliable when abstracted from the electronic medical record (e.g., a more detailed social history, establishing premorbid functional status, and independent confirmation of past medical history), and will require an informed consent process to allow the research team to approach subjects or their surrogates.

Similar databases exist at other centers for neurocritical care and have been central to the identification of characteristics, both predictive and associative, of patient outcomes. Done properly, this repository can facilitate many NCCU priorities including hypothesis generating, determining feasibility of single-site trials or involvement in multi-center trials, multimodal monitoring, biomarker research, quality improvement, and resident education.

All data will be collected from the patient medical record, patient bedside monitors, radiology PACS, and laboratory systems. The collection of data will not affect nor delay patient treatment at any instance.

Potential subjects will include patients admitted to University of Maryland's 22-bed NCCU for treatment of a life-threatening neurological illness. All patients 18 years of age and older will be eligible for participation in the study.

At the time study personnel approach the patient or the patient's surrogate to discuss the study, they will be provided with three options: (a) Full Consent, (b) Partial Refusal, or (c) Complete Refusal.

Subject's medical treatment will conform to existing clinical management protocols including routine ICU care. Standard ICU protocols call for assessments of mental status several times a day. The investigators would like to prospectively record the results of these exams in a rigorous, standardized manner. The investigators will attempt to correlate these assessments with clinical events and outcome. In addition to standard clinical treatment, details of each subject's hospitalization, demographic profile, past medical history, family history will be obtained by questionnaire and chart review. At discharge or 2 weeks after admission, a brief examination and mental status test will be performed. The subject and a family member or caregiver may also be asked to return for follow up evaluations 3 and 12 months after initial brain or spinal cord injury, in order to evaluate their longterm neurological status, disability, emotional status, cognitive functioning, and overall quality of life. These interviews may be conducted in person and will take approximately one hour each. For those patients unable to return in person, a shorter telephone interview will be conducted. Outcome measures may include the Glasgow Outcome Scale (GOS), the extended Glasgow Outcome Scale (eGOS), Modified Rankin Scale, Lawton Activities of Daily Living Index, Barthel Index, Sickness Impact Profile (SIP), NIH Stroke Scale, psychosocial assessments, memory and cognitive neuropsychometric tests (e.g. the Montreal Cognitive Assessment-MoCA).

Variables recorded during hospitalization will be examined for statistical correlation with neuropsychometric test results. Candidate pathophysiologic variables with independent predictive value for cognitive dysfunction, (e.g., including severity of illness upon admission, hydrocephalus, ischemia from vasospasm, and laboratory test results) will be identified using Pearson correlation and forward stepwise logistic regression. Relationships between acute pathology (e.g., lesions on neuroimaging or malignant electrical patterns on electroencephalography) and dysfunction within various cognitive domains (memory, attention, visuospatial ability, language) will be examined using contingency tables, Pearson correlation, linear regression, and the Wilcoxon signed rank test. If necessary, multivariate models will be used to confirm that significant independent relationships exist.

Blood samples will be analyzed to identify the factors causing secondary brain injury (e.g., the narrowing of the blood vessels (vasospasm) after initial hemorrhage).

For patients requiring an External Ventricular Drain (EVD) as part of their medical treatment, the cerebrospinal fluid (CSF) is drained into a collection bag, the amount of drainage recorded and the CSF discarded. The investigators may collect a 1 cc sample of the CSF daily prior to discard until it is medically warranted to remove the EVD or 14 days whichever comes first. NO EVD will be placed for the purposes of clinical research.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of potentially life-threatening neurological illness
* admitted to Neuro ICU within 14 days of initial injury

Exclusion Criteria:

* known pre-existing neurological deficits related to a developmental disorder
* prior severe stroke
* prior severe dementia
* prior severe head injury
* prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in University of Maryland Medical Center's Neurocritical Care Unit with potentially life-threatening neurological illness aged 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-09-08 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who score great than 60 on the Barthel Index | 3 month
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Scores range from 0 to 100. A higher score signifies better outcomes, more independent functionality.
Number of participants who score great than 26 on the Montreal Cognitive Assessment (MoCA) | 3 month
  The Montreal Cognitive Assessment was developed as a quick screening tool for neurological function. It assesses the domains of attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculation, and orientation. The MoCA has been tested extensively for use in a variety of disorders affecting cognition such as HIV, Huntington's chorea, Multiple Sclerosis, Parkinson's disease, stroke, vascular dementia, and substance abuse in addition to the wellness of older adults. The MoCA has been tested in ages ranging from as young as 49 in two reports to old-old (85+) with a variety of education levels. The total possible score is 30 points with a score of 26 or more considered normal.
Number of participants who score 1 or less on the Modified Rankin Scale | 3 month
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke. Scores range from 0 to 6. A lower score signifies better outcomes, more independent functionality.
Number of participants who have experienced adverse events | 3 month
  Medical history from hospital discharge to three months will help researchers learn of any adverse events or other medical complications.
Number of participants who score great than 75 on the EuroQOL | 3 month
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Y Parikh, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Zimmerman W, Pergakis M, Ahmad G, Morris NA, Podell J, Chang WT, Motta M, Chen H, Jindal G, Bodanapally U, Marc Simard J, Badjatia N, Parikh GY. Iodine-Based Dual-Energy Computed Tomography After Mechanical Thrombectomy Predicts Secondary Neurologic Decline from Cerebral Edema After Severe Stroke. Neurocrit Care. 2025 Jun;42(3):804-816. doi: 10.1007/s12028-024-02137-5. Epub 2024 Oct 24. PMID 39448427